CLINICAL TRIAL: NCT03685123
Title: Prescribed Exercise to Reduce Recidivism After Weight Loss Pilot (PREVAIL-P)
Brief Title: Exercise After Clinically Significant Weight Loss
Acronym: PREVAIL-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Collaborators: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Damon Swift, Assistant Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R56HL132961-01A1 (NIH)
Record Dates: First submitted 2018-09-22; First posted 2018-09-26 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Obesity; Sedentary Lifestyle; Insulin Resistance
Keywords: Exercise training; Insulin resistance; Lipids; Arterial stiffness; Fitness; Weight maintenance; Body composition; Energy expenditure; Weight loss
MeSH Terms: conditions — Obesity; Sedentary Behavior; Insulin Resistance; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PA-REC (Experimental): After achieving clinically significant weight loss, participants will exercise at the minimum physical activity recommendations
  Interventions: Behavioral: Physical activity recommendations
- WM-REC (Experimental): After achieving clinically significant weight loss, participants will exercise at the weight maintenance recommendations
  Interventions: Behavioral: Weight maintenance recommendations
- Weight Loss Phase (Experimental): All participant prior to randomization will undergo a weight loss phase. This will include weight loss with Optifast and supervised aerobic exercise training (2-3 times per week). The goal of participants are to lose 7% of body weight. After the weight loss phase, participants will be randomized to the study arms (PA-REC, WM-REC)
  Interventions: Behavioral: OPTIFAST weight loss

INTERVENTIONS:
Behavioral: Physical activity recommendations — Participants in the PA-REC group will exercise at 550 MET min. per week in a supervised format
  Arms: PA-REC
Behavioral: Weight maintenance recommendations — Participants in the WM-REC group will exercise at 970 MET min. per week in a supervised format
  Arms: WM-REC
Behavioral: OPTIFAST weight loss — Participants will participant in an OPTIFAST medical weight loss program and exercise training
  Arms: Weight Loss Phase

SUMMARY:
The Prescribed Exercise to Reduce Recidivism After Weight Loss Pilot (PREVAIL-P) study will evaluate the effect of aerobic exercise training amount on weight maintenance following clinically significant weight loss.

DETAILED DESCRIPTION:
The Prescribed Exercise to Reduce Recidivism After Weight Loss Pilot (PREVAIL-P) study will evaluate the effect of aerobic exercise training amount on weight maintenance following clinically significant weight loss (CWL). Overweight and obese (BMI: 25-40 kg/m2) men and women (18-65 years old) complete an OPTIFAST diet (7%-10% weight loss). Participants that obtain CWL will be subsequently randomized to aerobic exercise training consistent with the minimum physical activity guidelines (~150 min of moderate intensity exercise) or weight maintenance guidelines (200-300 min per wk. at moderate intensity) for 9 additional months.

Specific Aim 1: To demonstrate the efficacy of the weight loss program in producing CWL and retention/adherence of the exercise intervention. Overweight and obese adults (N=39) will participate in an OPTIFAST weight loss program and supervised aerobic exercise training (~550 metabolic equivalents minutes [MET min. per week.]) for 10 weeks. Participants who obtain CWL will be subsequently randomized to 16 weeks of aerobic training consistent with the minimum physical activity recommendations (~550 MET min per week.) or weight maintenance guidelines (~970 MET min per week). The percentage of participants that obtain at least 7% weight loss following OPTIFAST treatment, retention rates in the weight loss program, adherence to exercise levels, and changes in weight and cardiometabolic risk factors in response to the intervention will be evaluated.

Specific Aim 2: To test the hypothesis that exercise levels consistent with weight maintenance recommendations leads to greater weight maintenance after CWL compared to the minimum physical activity recommendation levels. Overweight and obese adults (N=30) enrolled in VIDANT health's OPTIFAST program and have achieved at least 7% weight loss will be randomized to 36 weeks of aerobic exercise training consistent with the minimum public health guidelines for physical activity (~550 MET min. per week.) or weight maintenance levels (~970 MET min per week). The effect of the intervention will be evaluated on weight (primary) as well as main secondary measures (e.g. body fat, visceral fat, lipids, lipoprotein particles size/class, insulin sensitivity, blood pressure, arterial stiffness, systemic inflammation, fitness, and quality of life). The aforementioned cardiometabolic risk factors were selected because they can be improved specifically by weight loss and thus may respond differently to weight maintenance or regain.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-65 years of age (postmenopausal females permitted)
* Body mass index: 25-39.9 kg/m2 at enrollment
* The capability and willingness to provide written informed consent
* Willingness to accept group assignment from randomization
* No resistance training and no structured aerobic exercise for > 20 minutes per day, 3+ days per week, for the last 6 months
* Conditions that are contraindicated for exercise training

Exclusion Criteria:

* Resting blood pressure > 180 mm Hg systolic and/or >100 mm Hg diastolic (individuals on blood pressure medications meeting the blood pressure criteria are eligible)
* Diagnosis of type 1 or 2 diabetes, and/or fasting glucose >125 mg/dL
* Medication for the treatment of type 1 or type 2 diabetes
* Bariatric surgery including gastric banding or bypass (potential effects on energy intake)
* Factors that may limit adherence to intervention or affect conduct of the trial
* Unable or unwilling to communicate with staff
* Failure to complete run-in or baseline testing
* Hospitalization for depression or severe mental illness in the last 6 months
* Not physically capable of performing the exercise required of the study protocol
* Consuming more than 14 alcoholic beverages per week
* Plan to be away from the Pitt County area more than 3 weeks in the next 3 months
* Lack support from a primary health care provider or family members
* Significant weight loss in the past year (> 20 pounds) or are currently using weight loss medications.
* Current diagnosis of schizophrenia, other psychotic disorders, or bipolar disorder
* Other temporary intervening event, such as sick spouse, or bereavement
* Other medical, psychiatric, or behavioral limitations that may interfere with study participation or the ability to follow the intervention protocol
* Underlying diseases or conditions likely to limit lifespan and/or affect the safety of the intervention
* Cancer requiring treatment in the past 5 years with anything but excellent prognosis
* Self-reported HIV, tuberculosis, Hepatitis B, or Hepatitis C
* History or evidence of serious arrhythmias, cardiomyopathy, congestive heart failure, aortic aneurism, myocardial infarction or heart transplantation
* Renal disease: urine protein > 100 mg/dl, serum creatinine ≥ 1.5 mg/dl or currently receiving dialysis.
* Auto-immune diseases (such as Lupus, Multiple Sclerosis, Graves' disease, or Rheumatoid arthritis)
* Chronic obstructive lung disease, peripheral vascular disease or angina that limits ability to follow exercise protocol
* History of stroke or transient ischemic attack
* History of vascular aneurysms
* History of bleeding disorders
* Pregnancy or plans to become pregnant
* Any other medical condition or disease that is life threatening or that can interfere with or be aggravated by exercise.
* Do not own smartphone for MyFitnessPal and Centrepoint Apps.
* Lack of an internet connection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Damon L Swift, Ph.D., Principal Investigator — East Carolina University
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prior to participants being randomized, they participated in a weight loss intervention. Thirty-nine participants were enrolled in that component of the trial as specified per protocol. Participants that obtained a weight loss goal of 7% were subsequently randomized to study groups. 36 participants completed the weight loss phase, and 33 of those individuals made the weight loss goal.
Pre-assignment Details: Participants have to make a weight loss goal in order to be assigned to be randomized in the present study. All participants completed an Optifast weight loss program after completing screening for inclusion/exclusion criteria. Participants that were able to obtain at least 7% weight loss were available for randomization in the present study
Groups:
- Weight Loss Phase: Prior to randomization into the groups, participants completed a weight loss phase. Only participants who were able to obtain 7% weight loss in the intervention proceeded to the study randomization groups (This is represented only in period 1 of this report)
- PA-REC: This group will participate in an OPTIFAST weight loss program. After achieving clinically significant weight loss, participants will exercise at the minimum physical activity recommendations
  Physical activity recommendations: Participants in the PA-REC group will exercise at 550 MET min. per week in a supervised format
  OPTIFAST weight loss: Participants will participant in an OPTIFAST medical weight loss program and exercise training
- WM-REC: This group will participate in an OPTIFAST weight loss program. After achieving clinically significant weight loss, participants will exercise at the weight maintenance recommendations
  Weight maintenance recommendations: Participants in the WM-REC group will exercise at 970 MET min. per week in a supervised format
  OPTIFAST weight loss: Participants will participant in an OPTIFAST medical weight loss program and exercise training
Period: Weight Loss Phase
Arm/Group | Weight Loss Phase | PA-REC | WM-REC
Started | 39 | 0 (Participants needed to achieve 7% weight loss to be randomized to study groups. Thus participants were randomized to this group after completion of the weight loss phase.) | 0 (Participants needed to achieve 7% weight loss to be randomized to study groups. Thus participants were randomized to this group after completion of the weight loss phase.)
Completed | 33 | 0 | 0
Not Completed | 6 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Did not obtain weight loss goal | 3 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — PI removal due to subject lack of compliance | 1 | 0 | 0
Period: Weight Maintenance Phase
Arm/Group | Weight Loss Phase | PA-REC | WM-REC
Started (After weight loss phase, participants are randomized to the PA-REC and the WM-REC. Thus there are no additional participant in the weight loss phase of this section.) | 0 (Weight loss phase is complete at this point in the study as participants are randomized to the PA-REC and WM-REC groups.) | 16 | 17
Completed | 0 | 12 | 9
Not Completed | 0 | 4 | 8
Not completed — Covid Pandemic | 0 | 4 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: This population is the baseline values for participants after the completion of the 10 week weight loss phase. Participants who met the weight loss goal of 7% were randomized to study groups.
Groups:
- Weight Loss Phase: All participants complete a weight loss phase prior to randomization to study groups. Participants participate in an optifast weight loss program where the goal is to lose 7% of their body weight. Participants who meet this goal are then randomized to the PA-REC or the WM-REC groups. (39 participants began the weight loss phase and 33 completed with 7% weight loss)
Arm/Group | Weight Loss Phase
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 13
  White | 23
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 39
Weight [Mean (Standard Deviation); unit: kilograms] | 95.0 (2.0)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 34.4 (0.6)
Body Fat perecntage [Mean (Standard Deviation); unit: Percent of total body composition] | 41.7 (0.9)
Lean Mass (kg) [Mean (Standard Deviation); unit: kg] | 53.6 (1.7)
Visceral fat mass [Mean (Standard Deviation); unit: grams] | 698.7 (33.5)
Absolute Fitness (unadjusted for body weight) [Mean (Standard Deviation); unit: L/min of oxygen consumption] — Fitness level quantified in liters per minute (not adjusted for body weight)
  L/min of oxygen consumption | 2.0 (0.1)
Relative Fitness (fitness adjusted by body weight) [Mean (Standard Deviation); unit: ml/kg/min of oxygen consumption] | 21.4 (0.7)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 117.0 (2.4)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 74.9 (1.7)
Glucose [Mean (Standard Deviation); unit: mg/dL] | 95.9 (1.5)
Insulin [Mean (Standard Deviation); unit: ulU/mL] | 16.6 (1.3)
LDL Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 114.3 (4.6)
HDL Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 52.4 (2.0)
Resting metabolic rate [Mean (Standard Deviation); unit: kcals/day] | 1545.2 (42.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: Weight will measured in a hospital gown on a balance beam scale. Change in weight will be calculated as the participant weight change from the end of the weight loss phase to the end of the weight maintenance phase (week 28 weight subtracted from the week 10 weight). A positive value indicates an increase in weight and a negative value indicates a reduction in weight
Time Frame: End of weight loss phase (week 10) to follow-up (week 28)
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | PA-REC | WM-REC
Number analyzed (Participants) | 12 | 9
kg | 0.7 (4.13) | -1.5 (4.65)
Statistical Analysis 1: Comparison: PA-REC vs WM-REC; Test type: Superiority; p = 0.256, Mixed Models Analysis

2. Secondary Outcome: Change in Cardiorespiratory Fitness
Description: Fitness will be measured using a modified Balke protocol on a treadmill. Participants will walk at an initial speed of 2.0 mph with 0% grade for the first 3 minutes after which the treadmill speed will increase to 3.0 mph for the next 3 minutes. The treadmill grade will be increased by 2.5% every 3 minutes until volitional exhaustion. Respiratory gases (VO2, CO2) and ventilation will be measured continuously using a True Max 2400 Metabolic Measurement Cart. Change in fitness will be quantified as the value at follow-up (week 28) subtracted from the value at week 10. An increase value will indicate an increase in fitness, while a decrease in the value will indicate a reduction in fitness
Time Frame: End of weight loss phase (week 10) to follow-up (week 28)
Measure: Mean (Standard Deviation); unit: L/min of oxygen consumption
Arm/Group | PA-REC | WM-REC
Number analyzed (Participants) | 12 | 9
L/min of oxygen consumption | 0.05 (0.094) | 0.16 (0.12)
Statistical Analysis 1: Comparison: PA-REC vs WM-REC; Test type: Superiority; p = 0.089, Mixed Models Analysis

3. Secondary Outcome: Change in Body Fat Percentage
Description: Dual-energy X-ray absorptiometry will be used to measure changes in fat mass and lean mass. Body fat will be quantified as the percent of fat relative to the total body mass. Lean mass will be quantified as the percent of lean tissue relative to the total body composition. This will be calculated at week 10 and at week 28. Change in these variables will be quantified as by subtracting the week 10 value from the week 28 value. Thus, a change in positive direction is associated with an increase in body fat or lean mass and a negative value represents a decrease.
Time Frame: End of weight loss phase (week 10) to follow-up (week 28)
Measure: Mean (Standard Deviation); unit: percentage of total body composition
Arm/Group | PA-REC | WM-REC
Number analyzed (Participants) | 12 | 9
percentage of total body composition | 0.89 (4.13) | -1.54 (2.3)
Statistical Analysis 1: Comparison: PA-REC vs WM-REC; Test type: Superiority; p = 0.244, Mixed Models Analysis

4. Secondary Outcome: Change in Waist Circumference
Description: Waist circumference will be measured at the natural waist (midway between the inferior border of the rib cage and the superior aspect of the iliac crest) with a gulick tape measure. Both landmarks (the inferior border of the ribcage and the superior aspect of the iliac crest) will be marked and the distance will be measured to determine the appropriate measurement site. Staff will confirm that: 1) the measurement tape remains horizontal; 2) the tape touches the entire circumference of the participant; 3) abdominal tissue is not compressed; 3) the tape measure is not within abdominal folds; 4) the measurement is taken at the end of normal respiration. The measurement will be repeated an additional time, and the reported value will be the average of these measurements. Both measurements must be within 0.5 cm to be considered acceptable for data purposes. The change in waist circumference will be quantified as the the week 28 value subtracted from the week 10 value.
Time Frame: End of weight loss phase (week 10) to follow-up (week 28)
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | PA-REC | WM-REC
Number analyzed (Participants) | 12 | 9
cm | 0.48 (3.1) | -2.4 (3.5)
Statistical Analysis 1: Comparison: PA-REC vs WM-REC; Test type: Superiority; p = 0.064, Mixed Models Analysis

5. Secondary Outcome: Changes in Blood Lipids Concentrations
Description: A fasting blood sample will be used to measure low density lipoprotein, high density lipoprotein, total cholesterol, and triglycerides will be measured. It will be quantified as the specific amount of the lipoprotein within the blood in mg/dL for all lipid variables. Participants will be fasted at least 12 hours prior to the blood draw. Change will be quantified as the week 28 value subtracted from the week 10 value. A positive value indicates an increase in the blood lipid variable and a negative value is associated with a reduction in the variable.
Time Frame: End of weight loss phase (week 10) to follow-up (week 28)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PA-REC | WM-REC
Number analyzed (Participants) | 12 | 9
mg/dL
  LDL cholesterol | 4.9 (18.7) | 5.4 (23.9)
  HDL cholesterol | 11.2 (10.7) | 7.5 (11.8)
  Total Cholesterol | 21.2 (14.7) | 15.5 (32.1)
  Triglycerides | 3.3 (15.5) | 13.1 (36.8)
Statistical Analysis 1: Comparison: PA-REC vs WM-REC; LDL levels; Test type: Superiority; p = 0.983, Mixed Models Analysis
Statistical Analysis 2: Comparison: PA-REC vs WM-REC; HDL levels; Test type: Superiority; p = 0.56, Mixed Models Analysis
Statistical Analysis 3: Comparison: PA-REC vs WM-REC; Total Cholesterol; Test type: Superiority; p = 0.71, Mixed Models Analysis
Statistical Analysis 4: Comparison: PA-REC vs WM-REC; Triglycerides; Test type: Superiority; p = 0.313, Mixed Models Analysis

6. Secondary Outcome: Change in Blood Pressure
Description: Brachial and aortic blood pressure will be measured using a sphygmocor XCEL. Blood pressure is quantified in mmHg and will be taken in the seated position after a 5 minute rest. Change in blood pressure is quantified by subtracting the week 28 value from the week 10 value. Thus, a positive number is associated with an increase in blood pressure across the time point and a decrease indicates a decrease in blood pressure
Time Frame: End of weight loss phase (week 10) to follow-up (week 28)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PA-REC | WM-REC
Number analyzed (Participants) | 12 | 9
mmHg
  Systolic blood pressure | 7.4 (9.6) | 9.2 (17.5)
  Diastolic blood pressure | 4.0 (5.9) | 6.37 (9.08)
  Aortic Systolic Blood Pressure | 6.6 (8.9) | 8.1 (14.6)
  Aortic diastolic blood pressure | 4.2 (6.4) | 6.1 (8.8)
Statistical Analysis 1: Comparison: PA-REC vs WM-REC; systolic Blood pressure; Test type: Superiority; p = 0.72, Mixed Models Analysis
Statistical Analysis 2: Comparison: PA-REC vs WM-REC; Diastolic Blood pressure; Test type: Superiority; p = 0.61, Mixed Models Analysis
Statistical Analysis 3: Comparison: PA-REC vs WM-REC; Change in aortic blood pressure between the PA-REC and the WM-REC Groups; Test type: Superiority; p = 0.1609, Mixed Models Analysis
Statistical Analysis 4: Comparison: PA-REC vs WM-REC; Change in aortic diastolic blood pressure between the PA-REC and WM-REC Groups; Test type: Superiority; p = 0.446, Mixed Models Analysis

7. Secondary Outcome: Change in Fasting Glucose Level
Description: Change in fasting glucose level. Fasting glucose level refers to the concentration of glucose within the blood (mg/dL). The change in fasting glucose level is quantified by subtracting the week 28 value from the week 10 value. Thus, a positive value indicates an increase in glucose level and a negative value indicates a decrease in glucose.
Time Frame: End of weight loss phase (week 10) to follow-up (week 28)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | PA-REC | WM-REC
Number analyzed (Participants) | 12 | 9
mg/dL | 2.1 (5.7) | 2.5 (6.4)
Statistical Analysis 1: Comparison: PA-REC vs WM-REC; Test type: Superiority; p = 0.965, Mixed Models Analysis

8. Secondary Outcome: Change in Fasting Insulin Level
Description: Fasting insulin represents the concentration of insulin in the blood. A positive value represents an increase in insulin concentration and a negative value represents a decrease in insulin concentration.
Time Frame: End of weight loss phase (week 10) to follow-up (week 28)
Measure: Mean (Standard Deviation); unit: ulU/mL
Arm/Group | PA-REC | WM-REC
Number analyzed (Participants) | 12 | 9
ulU/mL | 2.1 (5.48) | 178 (5.5)
Statistical Analysis 1: Comparison: PA-REC vs WM-REC; Test type: Superiority; p = 0.857, Mixed Models Analysis

9. Secondary Outcome: Change in Systemic Inflammation
Description: High sensitivity c-reactive protein is a marker of systemic inflammation and is quantified in mg/L. A postive value indicates an increase in c-reactive protein and a negative value represents a decrease in c-reactive protein.
Time Frame: End of weight loss phase (week 10) to follow-up (week 28)
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | PA-REC | WM-REC
Number analyzed (Participants) | 12 | 9
mg/L | -0.48 (0.78) | -0.43 (0.866)
Statistical Analysis 1: Comparison: PA-REC vs WM-REC; Test type: Superiority; p = 0.825, Mixed Models Analysis

10. Secondary Outcome: Change in Resting Metabolic Rate
Description: Resting metabolic rate (RMR) was measured in a quiet, temperature-controlled room using indirect calorimetry (TrueOne 2400, Parvo Medics, Salt Lake City, UT) with a clear ventilated canopy and dilution pump. Initially, participants rested in the seated position for 20 minutes. Participants then rested in the supine position in the dimly lit room for at least 20 additional minutes with the hood covering their head. RMR was determined from approximately 10 minutes of data at the end of the procedure when the FECO2 dilution was steadily maintained in the range of 1.0 and 1.2%. RMR data was considered valid when the coefficient of variations for resting energy expenditure, VO2 and VCO2, were ≤10% RMR will be expressed as the estimated amount of calories needed for a given a day (kcals/day). Change in RMR will be quantified as the week 28 value subtracted by the week 10 value. An increase in the value reflects an increase in RMR and a negative value represent a decrease.
Time Frame: End of weight loss phase (week 10) to follow-up (week 28)
Measure: Mean (Standard Deviation); unit: kcals per day
Arm/Group | PA-REC | WM-REC
Number analyzed (Participants) | 12 | 9
kcals per day | 75.2 (56.6) | -66.8 (65.4)
Statistical Analysis 1: Comparison: PA-REC vs WM-REC; Test type: Superiority; p = 0.061, Mixed Models Analysis

11. Secondary Outcome: Change in Insulin Sensitivity
Description: Insulin sensitivity will be measured using an oral glucose tolerance test. With the results of the oral glucose tolerance test at baseline, insulin sensitivity was calculated with the Matsuda index. Insulin sensitivity was calculated with Matsuda index: [10,000 / √glucose minute 0 x insulin minute 0) (mean glucose (OGTT) x mean insulin OGTT)]. A higher result is better.
Time Frame: End of Weight loss phase (week 10) to follow-up (week 28)
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | PA-REC | WM-REC
Number analyzed (Participants) | 12 | 9
Index | -1.16 (2.8) | -3.4 (11.0)

12. Secondary Outcome: Changes in Lipoprotein Size
Description: This measure describes the average size of the low density lipoprotein particles and high density lipoprotein participles
Time Frame: End of weight loss phase (week 10) to follow-up (week 28)
Measure: Mean (Standard Deviation); unit: nm
Arm/Group | PA-REC | WM-REC
Number analyzed (Participants) | 12 | 9
nm
  LDL Size | -0.04 (0.30) | 0.01 (0.27)
  HDL size | 0.21 (0.18) | 0.04 (0.30)
Statistical Analysis 1: Comparison: PA-REC vs WM-REC; Change in HDL particle size; Test type: Superiority — Change in particle size between the PA-REC and WM-REC groups; p = 0.105, Mixed Models Analysis
Statistical Analysis 2: Comparison: PA-REC vs WM-REC; Change in LDL particles; Test type: Superiority — Change in particle size between the PA-REC and the WM-REC groups; p = 0.849, Mixed Models Analysis

13. Secondary Outcome: Change in Arterial Stiffness (Pulse Wave Velocity)
Description: Arterial stiffness will be measured using pulse wave velocity. Participants will refrain from large meals and caffeine for at least 2 hours and alcohol, vigorous exercise and vasoactive medication for at least 12 hours. Testing will occur in a quiet temperature controlled room. Carotid to femoral pulse wave velocity (PWV) and aortic blood pressure parameters will be measured using a SphygmoCor XCEL (Itasca, IL). PWV will be obtained in the supine position after a 15-minute rest. Investigators will measure the speed of the pulse from the carotid (artery in neck) to the femoral artery (artery in the leg). PWV parameters will be obtained in duplicate in concert with current guidelines and will be quantified in m/sec.
Time Frame: End of weight loss phase (week 10) to follow-up (week 28)
Measure: Least Squares Mean (95% Confidence Interval); unit: m/sec
Arm/Group | PA-REC | WM-REC
Number analyzed (Participants) | 8 | 8
m/sec | 0.40 [-0.294934 to 1.108859] | 0.436787 [-0.265109 to 1.138684]

14. Secondary Outcome: Changes in Physical Activity Levels
Description: Participants will wear an ActivPal accelerometer for seven consecutive days, 24-hrs/day. The amount of time spent sitting and standing and steps will be calculated
Time Frame: Baseline to follow-up (week 28)
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | PA-REC | WM-REC
Number analyzed (Participants) | 12 | 9
steps per day | -437.02 (818.5) | 511.0 (2369.17)
Statistical Analysis 1: Comparison: PA-REC vs WM-REC; Change in steps per day from week 10 to week 28; Test type: Superiority; p = 0.278, ANOVA

15. Secondary Outcome: Change in Quality of Life: SF-36
Description: Quality of life (QOL) will be measured by the short form health survey (SF-36). SF36 consists of 36 questions that measure patient's HRQoL in 8 domains: physical functioning (PF), role-physical (RP), bodily pain (BP), general health (GH) that represent the physical HRQoL, vitality (VT), social functioning (SF), role-emotional (RE), and mental health (MH) that represent the mental HRQoL. Each domain is scored from 0 (worst health status) to 100 (best health status).
  The SF-36 also produces a measure of overall physical health (physical component score [PCS]) and overall mental health (mental component score [MCS]). Scoring of these items are standardized using means and standard deviations from the general US population. Aggregate PCS and MCS scores are standardized using a linear T-Score transformation to have a mean of 50 and a standard deviation of 10.
Time Frame: End of weight loss phase (week 10) to Follow-up (week 28)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PA-REC | WM-REC
Number analyzed (Participants) | 12 | 9
score on a scale
  SF-36 General Health (GH) | -2.7 (3.4) | -0.19 (1.6)
  SF-36 Physical Health (PH) | -0.2 (1.66) | 0.71 (1.41)
  SF-36 Role Physical (RP) | 0.45 (2.76) | 0.00 (0.0)
  SF-36 Bodily Pain (BP) | -5.2 (6.36) | -2.41 (4.49)
  SF-36 Vitality (VT) | -0.60 (6.53) | -2.21 (6.33)
  SF-36 Social Function (SF) | -1.0 (2.11) | -0.63 (1.77)
  SF-36 Mental Health (MH) | -1.31 (4.29) | 0.33 (8.08)
  SF-36 Role Emotional (RE) | -2.4 (5.2) | -0.44 (1.24)
  SF-36 Mental health | -1.61 (4.73) | -0.63 (4.88)
  SF-36 Physical | -1.48 (2.60) | -0.54 (2.88)
Statistical Analysis 1: Comparison: PA-REC vs WM-REC; Change in SF-36 General Health (GH); Test type: Superiority; p = 0.238, Mixed Models Analysis
Statistical Analysis 2: Comparison: PA-REC vs WM-REC; Change in SF-36 Physical health (PH); Test type: Superiority — Between groups analysis between the change in PA-REC Group vs. the WM-REC Group; p = 0.124, Mixed Models Analysis
Statistical Analysis 3: Comparison: PA-REC vs WM-REC; Change in SF-36 role physical; Test type: Superiority — Between groups analysis between the change in PA-REC Group vs. the WM-REC Group; p = 0.769, Mixed Models Analysis
Statistical Analysis 4: Comparison: PA-REC vs WM-REC; Change in SF-36 Bodily Pain; Test type: Superiority — Between groups analysis between the change in PA-REC Group vs. the WM-REC Group; p = 0.352, Mixed Models Analysis
Statistical Analysis 5: Comparison: PA-REC vs WM-REC; Change in SF-36 Vitality; Test type: Superiority — Between groups analysis between the change in PA-REC Group vs. the WM-REC Group; p = 0.898, Mixed Models Analysis
Statistical Analysis 6: Comparison: PA-REC vs WM-REC; Change in SF-36 social function; Test type: Superiority — Between groups analysis between the change in PA-REC Group vs. the WM-REC Group; p = 0.444, Mixed Models Analysis
Statistical Analysis 7: Comparison: PA-REC vs WM-REC; Change in SF-36 Mental Health; Test type: Superiority — Change between the PA-REC group and the WM-REC group; p = 0.537, Mixed Models Analysis
Statistical Analysis 8: Comparison: PA-REC vs WM-REC; Change in SF-36 Role Emotional; Test type: Superiority; p = 0.448, Mixed Models Analysis
Statistical Analysis 9: Comparison: PA-REC vs WM-REC; Change in SF-36 Mental Health (Sum); Test type: Superiority — Change between the PA-REC group and the WM-REC group; p = 0.537, Mixed Models Analysis
Statistical Analysis 10: Comparison: PA-REC vs WM-REC; Change in SF-36 Physical Health (sum); Test type: Superiority — Change between the PA-REC group and the WM-REC group; p = 0.482, Mixed Models Analysis

16. Secondary Outcome: Weight Loss Phase- Change in Dietary Composition
Description: Food Frequency Questionnaire (FFQ) contains approximately 105 items grouped by categories and is completed for both frequency of consumption as well as portion size selections by the individual. The questionnaire, upon completion, provides estimated daily intake values for selected nutrients (kilocalories, macronutrients, and micronutrients) and provides information on food group servings.
Time Frame: Baseline to follow-up (week 28)
Measure: Mean (Standard Deviation); unit: Kcals
Arm/Group | Weight Loss Phase
Number analyzed (Participants) | 36
Kcals | -1320.9 (169.7)

17. Other Pre Specified Outcome: Weight Loss Phase- Change in Weight (kg)
Description: The participants are weighed on scale in a hospital gown
Time Frame: Baseline to 10 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Weight Loss Phase
Number analyzed (Participants) | 36
kg | -8.8 (0.6)
Statistical Analysis 1: Comparison: Weight Loss Phase; Test type: Superiority; p < 0.001, Mixed Models Analysis

18. Other Pre Specified Outcome: Weight Loss Phase- Cardiorespiratory Fitness (L/Min)
Description: as for outcome 2
Time Frame: Baseline 0 to Week 10
Measure: Mean (Standard Deviation); unit: l/min
Arm/Group | Weight Loss Phase
Number analyzed (Participants) | 36
l/min | 2.0 (0.0)
Statistical Analysis 1: Comparison: Weight Loss Phase; Test type: Superiority; p = 0.37, Mixed Models Analysis

19. Other Pre Specified Outcome: Weight Loss Phase-Change in Body Fat (%)
Description: Dual-energy X-ray absorptiometry will be used to measure changes in fat mass and lean mass. Body fat will be quantified as the percent of fat relative to the total body composition. Lean mass will be quantified as the percent of lean tissue relative to the total body composition. Change in these variables will be quantified as by subtracting the week 10 value from the week 28 value. Thus, a change in positive direction is associated with an increase in body fat or lean mass and a negative value represent a decrease.
Time Frame: Baseline to Week (10)
Measure: Mean (Standard Deviation); unit: % body fat
Arm/Group | Weight Loss Phase
Number analyzed (Participants) | 36
% body fat | -2.1 (0.3)
Statistical Analysis 1: Comparison: Weight Loss Phase; Change in body fat; Test type: Superiority; p < 0.001, Mixed Models Analysis

20. Other Pre Specified Outcome: Weight Loss Phase- Change in Waist Circumference (cm)
Description: as for outcome 4
Time Frame: Baseline to Week 10
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Weight Loss Phase
Number analyzed (Participants) | 36
cm | -8.6 (0.8)
Statistical Analysis 1: Comparison: Weight Loss Phase; Test type: Superiority; p < 0.001, Mixed Models Analysis

21. Other Pre Specified Outcome: Weight Loss Phase-Changes in Blood Lipids Concentrations (mg/dL)
Description: A fasting blood sample will be used to measure low density lipoprotein, high density lipoprotein, total cholesterol, and triglycerides will be measured. It will be quantified as the specific amount of the lipoprotein within the blood in mg/dL for all lipid variables. Participants will be fasted at least 12 hours prior to the blood draw. Change will be quantified as the week 10 value subtracted from the week baseline value
Time Frame: Baseline to Week 10
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Weight Loss Phase
Number analyzed (Participants) | 36
mg/dL
  Low density lipoprotein (LDL) | -8.3 (2.7)
  High density lipoprotein (HDL) | -2.4 (1.1)
  Triglycerides | -24.1 (6.3)
  Total Cholesterol | -15.6 (3.2)
Statistical Analysis 1: Comparison: Weight Loss Phase; LDL; Test type: Superiority; p = 0.004, Mixed Models Analysis
Statistical Analysis 2: Comparison: Weight Loss Phase; Change in HDL; Test type: Superiority; p = 0.04, Mixed Models Analysis
Statistical Analysis 3: Comparison: Weight Loss Phase; Change in Total Cholesterol; Test type: Superiority; p < 0.001, Mixed Models Analysis
Statistical Analysis 4: Comparison: Weight Loss Phase; Triglycerides; Test type: Superiority; p < 0.001, Mixed Models Analysis

22. Other Pre Specified Outcome: Weight Loss Phase- Changes in Blood Pressure (mmHg)
Description: Brachial and aortic blood pressure will be measured using a sphygmocor XCEL. Blood pressure is quantified in mmHg and will be taken in the seated position after a 5 minute rest. Change in blood pressure is quantified by subtracting the week 10 value from the baseline value. Thus, a positive number is associated with an increase in blood pressure across the time point and a decrease indicates a decrease in blood pressure
Time Frame: Baseline to Week 10
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Weight Loss Phase
Number analyzed (Participants) | 36
mmHg
  Brachial systolic blood pressure | -6.8 (0.46)
  Brachial diastolic blood pressure | -5.9 (1.6)
  Aortic systolic blood pressure | -8.3 (8.9)
  Aortic diastolic blood pressure | -5.8 (6.3)
Statistical Analysis 1: Comparison: Weight Loss Phase; Test type: Superiority; p = 0.01, Mixed Models Analysis — Systolic blood pressure
Statistical Analysis 2: Comparison: Weight Loss Phase; Diastolic blood pressure; Test type: Superiority; p = 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Weight Loss Phase; Aortic blood pressure (mmHg); Test type: Superiority; p < 0.001, Mixed Models Analysis
Statistical Analysis 4: Comparison: Weight Loss Phase; Change in aortic diastolic pressure; Test type: Superiority; p < 0.001, Mixed Models Analysis

23. Other Pre Specified Outcome: Weight Loss Phase-Change in Blood Glucose
Description: Change in fasting glucose level. Fasting glucose level refers to the concentration of glucose within the blood (mg/dL). The change in fasting glucose level is quantified by subtracting the week 10 value from the baseline value. Thus, a positive value indicates an increase in glucose level and a negative value indicates a decrease in glucose.
Time Frame: Baseline to week 10
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Weight Loss Phase
Number analyzed (Participants) | 36
mg/dL | -11.0 (1.3)
Statistical Analysis 1: Comparison: Weight Loss Phase; Test type: Superiority; p < 0.001, Mixed Models Analysis

24. Other Pre Specified Outcome: Weight Loss Phase- Change in Insulin
Description: as for outcome 8
Time Frame: Baseline to Week 10
Measure: Mean (Standard Deviation); unit: (ulU/mL)
Arm/Group | Weight Loss Phase
Number analyzed (Participants) | 36
(ulU/mL) | -10.5 (1.1)
Statistical Analysis 1: Comparison: Weight Loss Phase; Test type: Superiority; p < 0.001, Mixed Models Analysis

25. Other Pre Specified Outcome: Weight Loss Phase-Change in Systemic Inflammation
Description: High sensitivity c-reactive protein is a marker of systemic inflammation and is quantified in mg/L. A positive value indicates an increase in c-reactive protein and a negative value represents a decrease in c-reactive protein.
Time Frame: Baseline to Week 10
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Weight Loss Phase
Number analyzed (Participants) | 36
mg/L | -0.3 (0.3)
Statistical Analysis 1: Comparison: Weight Loss Phase; Test type: Superiority; p = 0.366, Mixed Models Analysis

26. Other Pre Specified Outcome: Weight Loss Phase- Change in Resting Metabolic Rate
Description: Resting metabolic rate (RMR) was measured in a quiet, temperature-controlled room using indirect calorimetry (TrueOne 2400, Parvo Medics, Salt Lake City, UT) with a clear ventilated canopy and dilution pump. Initially, participants rested in the seated position for 20 minutes. Participants then rested in the supine position in the dimly lit room for at least 20 additional minutes with the hood covering their head. RMR was determined from approximately 10 minutes of data at the end of the procedure when the FECO2 dilution was steadily maintained in the range of 1.0 and 1.2%. RMR data was considered valid when the coefficient of variations for resting energy expenditure, VO2 and VCO2, were ≤10% RMR will be expressed as the estimated amount of calories needed for a given a day (kcals/day). Change in RMR will be quantified as the week 10 value subtracted by the baseline. An increase in the value reflects an increase in RMR and a negative value represent a decrease.
Time Frame: Baseline to Week 10
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Weight Loss Phase
Number analyzed (Participants) | 36
kcal/day | -111 (25.7)
Statistical Analysis 1: Comparison: Weight Loss Phase; Test type: Superiority; p < 0.001, Mixed Models Analysis

27. Other Pre Specified Outcome: Weight Loss Phase-Change in Insulin Sensitivity
Description: as for outcome 11
Time Frame: Baseline to Week 10
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Weight Loss Phase
Number analyzed (Participants) | 36
Index | 3.7 (0.9)

28. Other Pre Specified Outcome: Weight Loss Phase- Change in Augmentation Index
Description: Central Arterial stiffness will be measured using a SphygmoCor XCEL (Itasca, IL). Participants will refrain from large meals and caffeine for at least 2 hours and alcohol, vigorous exercise and vasoactive medication for at least 12 hours. Testing will occur in a quiet temperature controlled room in the seated position after a 5 minute rest. Augmentation index represent central arterial stiffness and will be quantified via augmentation index (%). The augmentation index (AIx) is a measure of systemic arterial stiffness, and is defined as the ratio of augmentation (Δ P) to central pulse pressure and expressed as percent. AIx = (ΔP/PP) x 100, where P = pressure and PP = Pulse Pressure. A lower value indicates better stiffness
Time Frame: Baseline to Week 10
Measure: Median (Standard Deviation); unit: Percent
Arm/Group | Weight Loss Phase
Number analyzed (Participants) | 34
Percent | -4.5 (1.5)
Statistical Analysis 1: Comparison: Weight Loss Phase; Test type: Superiority; p = 0.004, Mixed Models Analysis

29. Other Pre Specified Outcome: Weight Loss Phase- Change in Physical Activity Levels
Description: as for outcome 14
Time Frame: Baseline to Week 10
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Weight Loss Phase
Number analyzed (Participants) | 36
steps per day | 1562.4 (1890.3)
Statistical Analysis 1: Comparison: Weight Loss Phase; Test type: Superiority; p < 0.001, Mixed Models Analysis

30. Other Pre Specified Outcome: Weight Loss Phase- Change in Quality of Life: SF-36
Description: as for outcome 15
Time Frame: Baseline to Week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Weight Loss Phase
Number analyzed (Participants) | 36
score on a scale
  Global health | 4.6 (1.1)
  Physical Health | 5.3 (1.0)
  Role physical | 3.4 (1.4)
  Bodily Pain | 4.4 (1.0)
  Vitality | 6.6 (1.2)
  Social Functioning | 4.2 (1.2)
  Mental Health | 2.9 (1.1)
  Role Emotional | 5 (1.1)
  Mental health Components (Sum) | 4.0 (1.1)
  Physical health components (Sum) | 4.8 (1.2)
Statistical Analysis 1: Comparison: Weight Loss Phase; Test type: Superiority; p < 0.001, Mixed Models Analysis — General Health
Statistical Analysis 2: Comparison: Weight Loss Phase; Physical Health; Test type: Superiority; p < 0.001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Weight Loss Phase; Role physical; Test type: Superiority; p = 0.023, Mixed Models Analysis
Statistical Analysis 4: Comparison: Weight Loss Phase; Test type: Superiority; p < 0.001, Mixed Models Analysis — Bodily Pain
Statistical Analysis 5: Comparison: Weight Loss Phase; Vitality; Test type: Superiority; p < 0.001, Mixed Models Analysis
Statistical Analysis 6: Comparison: Weight Loss Phase; Social Functioning; Test type: Superiority; p < 0.001, Mixed Models Analysis
Statistical Analysis 7: Comparison: Weight Loss Phase; Mental Health; Test type: Superiority; p = 0.0105, Mixed Models Analysis
Statistical Analysis 8: Comparison: Weight Loss Phase; Role Emotional; Test type: Superiority; p < 0.001, Mixed Models Analysis
Statistical Analysis 9: Comparison: Weight Loss Phase; SF-36 mental health Components (sum); Test type: Superiority; p = 0.01, Mixed Models Analysis
Statistical Analysis 10: Comparison: Weight Loss Phase; Physical Health Components Sum; Test type: Superiority; p < 0.001, Mixed Models Analysis

31. Other Pre Specified Outcome: Weight Loss Phase-Change in Dietary Composition
Description: as for outcome 16
Time Frame: Baseline to Week 10
Measure: Mean (Standard Deviation); unit: kcals
Arm/Group | Weight Loss Phase
Number analyzed (Participants) | 36
kcals | -1320.9 (169)
Statistical Analysis 1: Comparison: Weight Loss Phase; Change in kilocalories consumed from baseline to week 10; Test type: Superiority; p < 0.001, Mixed Models Analysis

32. Other Pre Specified Outcome: Changes in Lipoprotein Class/Size
Description: LDL particle Size. This measure describes the average size of the Low density lipoprotein particles
Time Frame: Baseline to Week 10
Measure: Mean (Standard Deviation); unit: nm
Arm/Group | Weight Loss Phase
Number analyzed (Participants) | 36
nm
  LDL particle size | 0 (0)
  HDL particle size | -0.1 (0.0)
Statistical Analysis 1: Comparison: Weight Loss Phase; Change in LDL Particle Size; Test type: Superiority; p = 0.658, Mixed Models Analysis
Statistical Analysis 2: Comparison: Weight Loss Phase; HDL participle size; Test type: Superiority; p = 0.07, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Information on adverse events were collected over the entire research study (e.g. assessment measures, weight loss phase, weight maintenance phase). The weight loss phase of the intervention was 10 weeks. The weight maintenance phase (where participants were randomized to the PA-REC or WM-REC groups) lasted for 18 additional weeks.
Groups:
- Weight Loss Phase: OPTIFAST weight loss: Participants will participant in an OPTIFAST medical weight loss program and exercise training. The exercise training component of the PA-REDC
- PA-REC: After achieving clinically significant weight loss, participants will exercise at the minimum physical activity recommendations. Physical activity recommendations: Participants in the PA-REC group will exercise at 550 MET min. per week in a supervised format
- WM-REC: After achieving clinically significant weight loss, participants will exercise at the weight maintenance recommendations
  Weight maintenance recommendations: Participants in the WM-REC group will exercise at 970 MET min. per week in a supervised format
  OPTIFAST weight loss: Participants will participant in an OPTIFAST medical weight loss program and exercise training
Arm/Group | Weight Loss Phase | PA-REC | WM-REC
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 0/39 | 1/16 | 0/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Weight Loss Phase (N=39) | PA-REC (N=16) | WM-REC (N=17)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Participant felt nauseous during oral glucose tolerance test
Lightheadedness (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Participant felt lightheaded on the treadmill

LIMITATIONS AND CAVEATS:
Loss of participants due to the COVID-19 pandemic caused disenrollment of participants in the last cohort of the weight maintenance phase (e.g. shown in participant flow section). This may have limited our ability to detect significant differences between groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/23/NCT03685123/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/23/NCT03685123/ICF_001.pdf